CLINICAL TRIAL: NCT02298348
Title: NANT N2013-02 A Phase I Study of Sorafenib and Cyclophosphamide/Topotecan in Patients With Relapsed and Refractory Neuroblastoma
Brief Title: Sorafenib and Cyclophosphamide/Topotecan in Patients With Relapsed and Refractory Neuroblastoma
Acronym: N2013-02
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: New Approaches to Neuroblastoma Therapy Consortium (Other)
Collaborators: University of California, San Francisco (Other); Children's Hospital Los Angeles (Other); Lucile Packard Children's Hospital (Other); Children's Hospital Medical Center, Cincinnati (Other); University of Michigan (Other); Seattle Children's Hospital (Other); Dana-Farber Cancer Institute (Other); The Hospital for Sick Children (Other); Children's Healthcare of Atlanta (Other); University of Chicago (Other); Cook Children's Health Care System (Other); Children's Hospital Colorado (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NANT 2013-02
Record Dates: First submitted 2014-08-26; First posted 2014-11-21 (Estimated); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Neuroblastoma
Keywords: Neuroblastoma; NANT; Sorafenib; Relapse
MeSH Terms: conditions — Neuroblastoma; Recurrence | interventions — Sorafenib; Cyclophosphamide; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sorafenib and Cyclophosphamide/Topotecan (Other): Sorafenib and Cyclophosphamide/Topotecan with growth factor support.
  Interventions: Drug: Sorafenib; Drug: Cyclophosphamide; Drug: Topotecan

INTERVENTIONS:
Drug: Sorafenib — Sorafenib -100-200mg/m2/dose (dose escalation), Orally BID continuously Days 1 thru 28 Cyclophosphamide - 250 mg/m2/day IV x 5 days - day 1 thru day 5 Topotecan - 0.75 mg/m2/day IV x 5 days - day 1 thru day 5
  Other Names: SORAFENIB TOSYLATE; NEXAVARTM , BAY 54-9085
Drug: Cyclophosphamide — 250mg/m2/day IV x5 days (Day 1 through Day 5 of each course)
  Other Names: Cytoxan
Drug: Topotecan — 0.75mg/m2.day IV x5 days (Day 1 through Day 5 of each course)
  Other Names: SKF-104864,; Hycamtin®

SUMMARY:
This study will combine three drugs: sorafenib, cyclophosphamide and topotecan.

Adding sorafenib to cyclophosphamide and topotecan may increase the effectiveness of this combination. The investigators first need to find out the highest dose of sorafenib that can be given safely together with cyclophosphamide and topotecan. This is the first study to test giving these three drugs together and will help determine the highest dose of sorafenib that can safely be given together with cyclophosphamide and topotecan to patients with resistant/relapsed neuroblastoma.

DETAILED DESCRIPTION:
This study will combine three drugs: sorafenib, cyclophosphamide and topotecan.

This study involves the use of an experimental drug, called sorafenib. Sorafenib blocks the function of a protein that is important in the growth of cancer cells. This drug has been tested by itself (as a single-agent) in children with relapsed solid tumors, including patients with neuroblastoma. In the laboratory, sorafenib appears to make neuroblastoma tumors smaller, and in addition can help immune cells to be more active in attacking tumors and blocks other harmful immune cells from promoting tumor growth and function. Sorafenib also helps to block tumor cells from developing blood vessels used to "feed" to tumor. Sorafenib is an FDA-approved drug currently widely used for adults with specific types of liver and kidney cancer.

Cyclophosphamide and topotecan are both FDA-approved chemotherapy drugs. These drugs are approved for the treatment of certain adult cancers, but have also been used to treat children with cancer. These drugs have been used in combination in many people with neuroblastoma. In some neuroblastoma patients, this combination has reduced the amount of tumor burden.

Adding sorafenib to cyclophosphamide and topotecan may increase the effectiveness of this combination. The investigators first need to find out the highest dose of sorafenib that can be given safely together with cyclophosphamide and topotecan. This is the first study to test giving these three drugs together and will help determine the highest dose of sorafenib that can safely be given together with cyclophosphamide and topotecan to patients with resistant/relapsed neuroblastoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be < 30 years of age when registered on study.
* Patients must have a diagnosis of neuroblastoma either by histologic verification of neuroblastoma and/or demonstration of tumor cells in the bone marrow with increased urinary catecholamines.
* Patients must have high-risk neuroblastoma according to COG risk classification at the time of study enrollment. Patients who were initially considered low or intermediate risk, but then reclassified as high risk are also eligible.
* Patients must have at least ONE of the following:

Recurrent/progressive disease at any time prior to study enrollment - regardless of response to frontline therapy.

Refractory disease: persistent sites of disease after achieving a best overall response of no response to front line therapy after a minimum of 4 cycles of induction therapy AND patient has never had recurrent/progressive disease.

Persistent disease: persistent sites of disease after achieving a best overall response of partial response to frontline therapy after a minimum of 4 cycles of induction therapy AND patient has never had recurrent/progressive disease.

* Patients must have at least ONE of the following (lesions may have received prior radiation therapy as long as they meet the other criteria listed below):
* At least one MIBG avid bone site or diffuse MIBG uptake.

  * For recurrent/progressive or refractory disease, a biopsy is not required regardless of number of MIBG avid lesions
  * For persistent disease, if patient has only 1 or 2 MIBG avid lesions OR a Curie core of 1 - 2, then biopsy confirmation of neuroblastoma and/or ganglioneuroma in at least one site present at the time of enrollment (bone marrow, bone or soft tissue) is required to be obtained at any time point prior to enrollment and two weeks subsequent to most recent prior therapy. If a patient has 3 or more MIBG avid lesions OR a Curie Score of ≥ 3 then no biopsy is required for eligibility.
* Any amount of neuroblastoma tumor cells in the bone marrow based on routine morphology (with or without immunocytochemistry) in at least one sample from bilateral aspirates and biopsies.
* At least one soft tissue site that meets criteria for a TARGET lesion defined by:

  * Size: Lesion can be accurately measured in at least one dimension with a longest diameter ≥ 10mm, or for lymph nodes ≥ 15mm short axis. Lesions meeting size criteria will be considered measurable.
  * In addition to size, a site needs to meet one of the following criteria:

MIBG avid. For patients with persistent disease only: If a patient has only 1 or 2 MIBG avid lesions OR a Curie Score of 1 - 2, then biopsy confirmation of neuroblastoma and/or ganglioneuroblastoma in at least one site present at time of enrollment (either bone marrow, bone and/or soft tissue) is required to be obtained at any time point prior to enrollment and at least two weeks subsequent to most recent prior therapy. If a patient has 3 or more MIBG avid lesions OR a Curie Score of ≥ 3 then no biopsy is required for eligibility.

* FDG-PET avid (only if tumor known to be MIBG non-avid). These patients must have had a biopsy confirming neuroblastoma and/or ganglioneuroblastoma in at least one FDG-PET avid site present at the time of enrollment done prior to enrollment and at least two weeks subsequent to the most recent prior therapy.
* Non-avid lesion (both MIBG and FDG-PET non-avid). These patients must have had a biopsy confirming neuroblastoma and/or ganglioneuroblastoma in at least one non-avid lesion present at the time of enrollment done prior to enrollment and at least two weeks subsequent to the most recent prior therapy.
* Patients must have a life expectancy of at least 8 weeks and a Lansky (< 16 years age) or Karnofsky (> 16 years age) score of at least 50
* Patients must have fully recovered from the acute toxic effects of all previous chemotherapy, immunotherapy, or radiotherapy prior to study enrollment.
* Patients must not have received the therapies indicated below for the specified time period prior to the first day of administration of protocol therapy on this study:
* Myelosuppressive chemotherapy: Last dose was given at least 14 days before the start date for protocol therapy.
* Biologic (anti-neoplastic agent including retinoids): Last dose given at least 7 days prior to the start date for protocol therapy.
* Monoclonal antibodies: Last dose of any monoclonal antibodies must have received at least 7 days or 3 half-lives, whichever is longer, prior to the start date for protocol therapy. Please refer to table posted at www.nant.org for definition of half-lives for specific monoclonal antibodies.
* Patients must not have received radiation for a minimum of two weeks prior to study enrollment.
* Patients are eligible 12 weeks after date of autologous hematopoietic stem cell infusion following myeloablative therapy (timed from first day of this protocol therapy).
* Patients are not eligible post allogeneic stem cell transplant.
* Patients who have received an autologous hematopoietic stem cell infusion to support non-myeloablative therapy (such as 131I-MIBG) are eligible at any time as long as they meet the other criteria for eligibility.
* A minimum of 6 weeks must have elapsed after 131I-MIBG therapy prior to start of protocol therapy.
* Patients who have received prior treatment with cyclophosphamide and topotecan are eligible if they did not have tumor relapse/progression while receiving this combination.
* Patients who have received prior treatment with sorafenib are eligible, as long as the sorafenib was not given in combination with cyclosphosphamide and/or topotecan. Patients with tumor relapse/progression while on sorafinib or having dose modifications or experiencing toxicity that required sorafenib to be discontinued are also ineligible to participate in this study.
* Growth factors that support platelet or white cell number or function must not have been administered within 7 days of blood draw documenting hematopoietic function (ANC, Platelets) eligibility. .
* Patients must not be receiving any other anti-cancer agents or radiotherapy at the time of study entry or while on study.
* Patients must not be receiving other investigational medications (covered under another IND) while on study.
* Treatment with clinically significant enzyme inducers, such as the enzyme-inducing antiepileptic drugs phenytoin, carbamazepine or phenobarbital, or rifampin, rifabutin, rifapentine or St. John's wort within 14 days prior to the first dose of sorafenib and during protocol therapy must not be used as these may interfere with sorafenib metabolism. Non-enzyme inducing anticonvulsants (Keppra, etc.) can be used after discussion with study chair.
* Patients must not be receiving active anti-coagulation therapy at the time of study entry (or while on study).
* Patients with cardiac arrhythmias must not be receiving anti-arrhythmic medication at time of study entry (or while on study).
* Patients must not be receiving anti-hypertensive medications at time of study entry.
* ANC: 1000/ul (no short acting hematopoietic growth factors within 7 7 days of blood draw documenting eligibility and no long-acting hematopoietic growth factors within 14 days of blood draw documenting eligibility)
* Platelet count: 100,000/ul and transfusion independent (no platelet transfusions within 7 days of blood draw documenting eligibility)
* Patients with known bone marrow metastatic disease will be eligible for study as long as they meet hematologic function criteria above.
* Hematuria ≤ 1+ on urinalysis
* Age-adjusted serum creatinine 1.5 x normal for age/gender
* Total bilirubin 1.5 x normal for age, AND
* SGPT (ALT) ≤ 135 U/L and SGOT (AST) ≤ 3X ULN. (for the purpose of this study, the upper limit of normal [ULN] for SGPT [ALT] is 45 U/L).
* Serum albumin > 2.5 g/dl
* Patient must have blood pressure ≤ 95th percentile for age, height, and gender
* Patients may not be on medical therapy for hypertension at time of enrollment.
* Patient must have a QT/QTc interval ≤ 450 msec.
* INR and aPTT < 1.2 times upper limit of normal for age.
* No history of bleeding diathesis.
* Amylase and Lipase < 1.5 x normal for age.
* Patients with other ongoing serious medical issues must be approved by the study chair prior to registration.

Exclusion Criteria:

* Subjects with calculated BSA < 0.40 m2 are not eligible for study participation as Sorafenib dosing for this study cannot accommodate subjects of this size utilizing commercially available drug formulation.
* Pregnancy: Serum B-HCG must be negative in girls who are post-menarchal. Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.
* Pregnant or breast-feeding women will not be entered on this study due to risks of fetal and teratogenic adverse events.
* Patients who have an active or uncontrolled infection are excluded. Patients on prolonged antifungal therapy are still eligible if they are culture and biopsy negative in suspected radiographic lesions and meet other organ function criteria.
* Patients with prior allogeneic transplant are not eligible.Patients with a documented history of cerebrovascular accidents and/or TIA within the past 6 months are not eligible.
* Patients with a history of intracranial hemorrhage are not eligible.
* Patients with a history of venous or arterial thrombosis personally or in a first degree relative before the age of 40 years are not eligible unless the thrombotic event was associated with a central line.
* Patient with prolonged QT/QTc (defined as QTc interval > 450 msec) are not eligible.
* Patient declines participation in NANT 04-05. (Neuroblastoma Biology Study)

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Estimated)
Dates: Start 2015-10-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The maximum tolerated dose of sorafenib given twice each day when given in combination with cyclophosphamide/topotecan for 5 days | 2 years
  By dose level (Dose Escalation of Sorafenib Only; The entry dose of sorafenib at 125 mg/m2 /dose is equivalent to 62.5% of the single agent MTD for pediatric solid tumor patients). Two to six evaluable patients will be entered at each of the three dose levels for determination of the maximum tolerated dose. The minimum sample size required to identify the MTD is 4 patients.
The number and types of toxicities of sorafenib when administered in combination with cyclophosphamide and topotecan. | 2 years
  Patients will be evaluable for inclusion in dose escalation consideration if they have received >80% of the 70 planned doses of sorafenib, >= 4 of the 5 planned doses of cyclophosphamide, and >=4 of the 5 planned doses of topotecan in course 1 AND are followed until Day 35 of the first course of therapy. In addition, patients who experience DLT at any time after the first dose of sorafenib are evaluable for inclusion in dose escalation consideration. Toxicity will be assessed and reported on all patients who begin sorafenib therapy. All toxicities observed will be summarized and graded using the CTCAE criteria, version 4.0 which can be downloaded from the CTEP home page (http://ctep.cancer.gov). The type of toxicities (organ affected or laboratory determination), severity, duration, and reversibility or outcome will be recorded. Toxicities observed during the first course of therapy (day -6 through day 28) will be assessed to define the MTD and guide dose escalation.

CONTACTS AND LOCATIONS:
Locations (12):
- United States (11):
  - Children's Hospital Los Angeles, Los Angeles, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Children Hospital of Colorado, Aurora, Colorado
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - University of Chicago, Comer Children's Hospital, Chicago, Illinois
  - Childrens Hospital Boston, Dana-Farber Cancer Institute., Boston, Massachusetts
  - C.S Mott Children's Hospital, Ann Arbor, Michigan
  - University of North Carolina, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cook Children's Healthcare System, Fort Worth, Texas
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
- Hospital for Sick Children, Toronto, Ontario, Canada